CLINICAL TRIAL: NCT04463368
Title: SCANDIUM II Trial - A Phase I Randomized Controlled Multicentre Trial of Isolated Hepatic Perfusion in Combination With Ipilimumab and Nivolumab in Patients With Uveal Melanoma Metastases
Brief Title: Isolated Hepatic Perfusion in Combination With Ipilimumab and Nivolumab in Patients With Uveal Melanoma Metastases
Acronym: SCANDIUM II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-587
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Uveal Melanoma; Liver Metastases
MeSH Terms: conditions — Uveal Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Patients will be treated with IHP followed by 4 courses of ipilimumab 3mg/kg and nivolumab 1mg/kg every third week followed by continued nivolumab 480mg q4w up to 1 year.
  Interventions: Procedure: Isolated hepatic perfusion; Drug: Ipilimumab; Drug: Nivolumab
- Arm B (Experimental): Patients will be treated with 1 course of ipilimumab 3mg/kg and nivolumab 1mg/kg followed by IHP after 3 weeks and then another 3 courses of ipilimumab 3mg/kg and nivolumab 1mg/kg every third week followed by continued nivolumab 480mg q4w up to 1 year.
  Interventions: Procedure: Isolated hepatic perfusion; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Procedure: Isolated hepatic perfusion — The procedure is performed under general anaesthesia. The caval vein is isolated infrahepatically above the renal veins and suprahepatically between the diaphragm and the pericardium. A catheter is placed in the retrohepatic portion of the caval vein for perfusion outflow. The portal vein is clamped and the proper hepatic artery is cannulated via the gastroduodenal artery. The liver perfusion is performed at a rate of 8- 9 ml/kg/min with a target liver temperature of 40 degrees Celsius. The leakage from the system was continuously recorded using Technetium labelled albumin (Vasculosis) injected into the perfusion circuit. Melphalan (1 mg/kg bodyweight divided into two doses, given 30 minutes apart) is added to the perfusion system. The perfusion is then continued for 60 minutes, after which the perfusion was discontinued.
Drug: Ipilimumab — 4 courses of ipilimumab 3mg/kg every third week
Drug: Nivolumab — 4 courses of nivolumab 1mg/kg every third week

SUMMARY:
Uveal melanoma is the most common primary intraocular malignancy in adults. Despite successful control of the primary tumour, metastatic disease will develop in approximately 35%-50% of the patients within 10 years. The liver is the most common site for metastases, and about 50% of the patients will have isolated liver metastases. Isolated hepatic perfusion is a regional treatment where the liver is completely isolated from the systemic circulation, allowing a high concentration of chemotherapy to be perfused through the liver with minimal systemic exposure. The introduction of modern immunotherapy in the treatment arsenal for cutaneous melanoma also creates hope for patients with uveal melanoma metastases. However, the results of immunotherapy have so far been disappointing. The reason for the low efficacy could be that uveal melanoma develops in the immune privileged eye.

The hypothesis in this trial is that isolated hepatic perfusion with melphalan causes an immunogenic type of cell death by local tumour destruction while leaving the immune-system intact. This will cause an activation of the immune-system and the addition of ipilimumab and nivolumab will enhance this effect, ultimately increasing the treatment efficacy.

The primary objective of this trial is to evaluate the safety and tolerability of isolated hepatic perfusion together with ipilimumab and nivolumab when given at the same time or as a sequenced regimen. The study design is a phase I randomized controlled, multicentre, open-label trial. Active follow-up will be performed for 2 years. Patients will be randomized after diagnoses of metastatic disease to one of the following treatment arms:

Arm A. Patients will be treated with IHP followed by 4 courses of ipilimumab 3mg/kg and nivolumab 1mg/kg every third week followed by continued nivolumab 480mg q4w up to 1 year.

Arm B. Patients will be treated with 1 course of ipilimumab 3mg/kg and nivolumab 1mg/kg followed by IHP after 3 weeks and then another 3 courses of ipilimumab 3mg/kg and nivolumab 1mg/kg every third week followed by continued nivolumab 480mg q4w up to 1 year.

ELIGIBILITY:
Inclusion Criteria

1. Patient is ≥18 years of age on the day of signing informed consent
2. Patient is willing and able to provide written informed consent and comply with study procedures. Written informed consent must be signed and dated before the start of specific protocol procedures
3. Patient must have a histologically confirmed diagnosis of stage IV uveal melanoma. If tissue biopsy is judged not feasible by the investigator, cytological diagnosis from fine needle aspiration (FNA) will be accepted
4. Measurable disease by computed tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria with at least one target lesion identified in the liver.
5. ECOG performance status of 0 or 1
6. No previous immunotherapy for uveal melanoma metastases.
7. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
8. Female patients of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
9. Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria

1. Life expectancy of less than 3 months
2. Body mass index above 35
3. More than 50% of the liver volume replaced by tumor as measured by CT or MRI
4. Known congestive heart failure with an LVEF <40%
5. COPD or other chronic pulmonary disease with PFT's indicating an FEV< 50% predicted for age
6. Interstitial lung disease (ILD) or (non-infectious) pneumonitis
7. Reduced renal function defined as S-Creatinine >=1.5xULN or Creatinine Clearance < 40 mL/min, calculated using the Cockroft and Gault formula
8. Reduced hepatic function (defined as AST, ALT, bilirubin>3*ULN and PK-INR>1.5) or medical history of liver cirrhosis or portal hypertension
9. Hemoglobin <90 g/L or platelets <100x109/L or neutrophils <1.5x109/L
10. Use of live vaccines four weeks before or after the last study treatment
11. History of severe hypersensitivity reactions to mAbs
12. Known human immunodeficiency virus (HIV) infection, acquired immunodeficiency syndrome (AIDS), hepatitis B or hepatitis C
13. Active autoimmune disease or a history of known or suspected autoimmune disease
14. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
15. Concomitant therapy with any other anti-cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications or use of other investigational drugs
16. Has a known additional malignancy that is progressing or requires active treatment.
17. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.
18. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 1 year
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Evaluation of objective response rate (ORR)
Clinical benefit rate (CBR) | 2 years
  Evaluation of clinical benefit rate (CBR)
Progression-free survival (PFS) | 2 years
  Evaluation of progression-free survival (PFS)
Hepatic progression-free survival (hPFS) | 2 years
  Evaluation of hepatic progression-free survival (hPFS)
Overall survival (OS) | 2 years
  Evaluation of overall survival (OS)
Time to response (TTR) | 2 years
  Evaluation of time to response (TTR)
Duration of response (DOR) | 2 years
  Evaluation of duration of response (DOR)

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided